CLINICAL TRIAL: NCT03326882
Title: Comparison of Glidescope Videolaryngoscope and Macintosh Laryngoscope in Children Aged >1 Years
Brief Title: Glidescope Videolaryngoscope and Macintosh Laryngoscope in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sisli Hamidiye Etfal Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Canan Tulay ISIL, M.D., Sisli Hamidiye Etfal Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: SEEAH
Record Dates: First submitted 2017-10-24; First posted 2017-10-31 (Actual); Last update posted 2017-10-31 (Actual); Status verified 2017-10

CONDITIONS: Anesthesiology; Pediatrics
MeSH Terms: interventions — Intubation, Intratracheal

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Glidescope (Active Comparator): A device for endotracheal intubation
  Interventions: Device: Endotracheal intubation
- Macintosh laringoscope (Active Comparator): A device for endotracheal intubation
  Interventions: Device: Endotracheal intubation

INTERVENTIONS:
Device: Endotracheal intubation
  Other Names: Glidescope video laryngoscope

SUMMARY:
The main objective of this study was to evaluate the intubation time of Glidescope compared with Macintoch laryngoscope in pediatric patients, ease of intubation, and cardiovascular changes during intubation.

DETAILED DESCRIPTION:
This was a prospective randomized clinical study to be performed in pediatric patients older than 1 years who are undergoing surgical procedures requiring endotracheal intubation. Time to endotracheal intubation was compared between patients intubated using a GlideScope® video laryngoscope, and those intubated by standard direct laryngoscopy. The main objective of this study was to evaluate the intubation time of Glidescope compared with Macintoch laryngoscope in pediatric patients, ease of intubation, and cardiovascular changes during intubation.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status I-II patients,
* scheduled for elective surgery under general anesthesia with endotracheal intubation

Exclusion Criteria:

* risk of pulmonary aspiration,
* presence of difficult intubation,
* emergency surgery,
* cardiovascular disease,
* respiratuar disease,
* hemodynamic instability.

Ages: 1 Year to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2016-02; Primary Completion 2016-03 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Duration of Intubation | Intraoperative
  Time from laryngoscopy to intubation

CONTACTS AND LOCATIONS:
Overall Officials: Canan Tulay Isil, Study Director — Sisli Hamidiye Etfal Training and Research Hospital

IPD SHARING:
Plan to Share IPD: No
This kind of data can only be shared with additional governemental agreement.

REFERENCES:
- [Background] Holm-Knudsen RJ, Rasmussen LS. Paediatric airway management: basic aspects. Acta Anaesthesiol Scand. 2009 Jan;53(1):1-9. doi: 10.1111/j.1399-6576.2008.01794.x. PMID 19128325